CLINICAL TRIAL: NCT03596788
Title: Effects of Different Sports Supplements on Metabolism and Perceptual Responses During Distance Running
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Assistant Professor, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1223706-2
Record Dates: First submitted 2018-06-28; First posted 2018-07-24 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Anomalies Gastrointestinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbohydrate Beverage (Experimental): A glucose-fructose beverage mixture supplying 100 grams of carbohydrate per day for 5 days
  Interventions: Dietary Supplement: Carbohydrate Beverage
- Placebo Beverage (Placebo Comparator): An artificially-sweetened beverage containing aspartame
  Interventions: Dietary Supplement: Placebo Beverage

INTERVENTIONS:
Dietary Supplement: Carbohydrate Beverage — The carbohydrate beverage will supply approximately 100 grams of carbohydrate per day (in the form of glucose and fructose)
  Arms: Carbohydrate Beverage
Dietary Supplement: Placebo Beverage — The placebo beverage will contain aspartame.
  Arms: Placebo Beverage

SUMMARY:
Several previous studies have shown that repeatedly ingesting carbohydrate supplements during exercise training sessions, over a period of days and weeks, can gradually increase carbohydrate oxidation and reduce gut discomfort during exercise. However, repeatedly ingesting large amounts of carbohydrate during training sessions can be burdensome and can cause gut distress. Thus, it would be advantageous if the same long-term benefits could be realized from consuming these carbohydrate supplements at rest instead of specifically during training sessions. Therefore, the goal of this study is to examine whether repeatedly ingesting a carbohydrate-rich beverage at rest over a 5-day period alters metabolism and gut symptoms while ingesting carbohydrate during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Be currently running ≥15 miles per week
* Have completed at least one run >60 minutes over the past month
* Have completed one or more marathons within the past year

Exclusion Criteria:

* Overt cardiovascular disease or metabolic disorder
* Adverse symptoms (e.g., unusual shortness of breath, dizziness, chest pain) with exercise
* Allergies/intolerances to any of the ingredients in the beverages

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Ratings | Symptoms will be collected during a 60 minute run on a treadmill at a baseline visit and at a second visit after ingesting the carbohydrate or placebo beverage for 5 days.
  Symptoms such as nausea, fullness, belching, reflux, abdominal cramps, flatulence, and urge to defecate will be recorded on a 0-10 scale (0 = no discomfort, 10 = unbearable discomfort).
Change in Hydrogen Breath Production | Samples will be collected before after a 60-minute run at a baseline visit and at a second visit after ingesting the carbohydrate or placebo beverage for 5 days.
  Samples of expired air will be tested for hydrogen levels, a marker of carbohydrate malabsorption

SECONDARY OUTCOMES:
Change in Carbohydrate Oxidation | Respiratory gases will be collected during each 60-minute run at a baseline visit and at a second visit after ingesting the carbohydrate or placebo beverage for 5 days.
  Respiratory gases will be used to estimate carbohydrate oxidation rates.
Change in Feeling Scale | Ratings will be collected collected before and during each 60-minute run at a baseline visit and at a second visit after ingesting the carbohydrate or placebo beverage for 5 days.
  A bipolar scale ranging from -5 (very bad) to +5 (very good)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wilson, PhD, Principal Investigator — Old Dominion University
Locations (1):
- Human Performance Lab, Norfolk, Virginia, United States